CLINICAL TRIAL: NCT04561882
Title: Transcatheter Exclusion of Atrial Septal Aneurysm Via Transseptal Perforation: First-in-human Use Study
Brief Title: Transcatheter Exclusion of Atrial-septal-aneurysm (TEA)
Acronym: TEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-7
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Atrial Septal Aneurysm
Keywords: atrial septal aneurysm; patent foramen ovale; defect; stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter exclusion of atrial septal aneurysm (Experimental): Transcatheter reconstruction of atrial septum might be achieved with PFO occluder through transseptal perforation in patients with ASA.
  Interventions: Device: Transcatheter exclusion of atrial septal aneurysm

INTERVENTIONS:
Device: Transcatheter exclusion of atrial septal aneurysm — Through transseptal perforation, transcatheter reconstruction of atrial septum was achieved with PFO occluder to cover the whole ASA.
  Device: Cardi-O-Fix™ patent foramen ovale occluder (Starway Medical Technology, Inc. Beijing, CN)

SUMMARY:
This study aims to investigate the safety and efficacy of transcatheter exclusion of atrial septal aneurysm (ASA) via transseptal perforation in patients with ASA.

DETAILED DESCRIPTION:
Atrial septal aneurysm (ASA) has been considered a potential cardiac source of embolism, and its prevalence is about 1%. In adult patients with stroke and normal carotid arteries, ASA is an important predictor of recurrent stroke. The most common abnormalities associated are interatrial shunts, that is, a patent foramen ovale (PFO) or an atrial septal defect (ASD). For large ASA with interatrial shunt, it is difficult to cover ASA with conventional devices, which might result in unstability of occluders and related complications . For isolated ASA with high risk, thrombus and emboli have been reported and anticoagulation has been used empirically.

In addition, the left atrial septal pouch can be considered as a special subtype of atrial septal aneurysm, in which thrombus might arise from the cavity of the pouch. Pervious researches have noted that left atrial septal pouch was a site of origin of thrombus formation and a source of embolism, and it was associated with cryptogenic stroke. For patients with ASA, we hypothesizes that transcatheter reconstruction of atrial septum might be achieved with PFO occluder through transseptal perforation. The aim of this study is to investigate the safety and efficacy of transcatheter exclusion of ASA via transseptal perforation.

This study will enroll subjects with ASA (including left atrial septal pouch), and enrollment will be divided into three phases.

Phase 1: large ASA patients with interatrial communication (ASD or PFO). A maximum of 30 patients is reached.

Phase 2: ASA patients with intact septum and high risk of cryptogenic stroke. A maximum of 20 patients is reached.

Phase 3: left atrial septal pouch with high risk of cryptogenic stroke. A maximum of 20 patients is reached.

ELIGIBILITY:
Inclusion Criteria:

1. In large-ASA patients with PFO (Phase1) (1)The length of ASA >20 mm and bulging >10 mm or a combined total excursion right and left > 15 mm; (2)Presence of a PFO indicated for device closure (Echocardiographic and/or transcranial Doppler evidence of right to left shunt at the atrial level); (3)History of cryptogenic stroke/TIA/migraine without other risks; (4) Failure to cover ASA after trial device-closure of PFO and the unstable device confirmed with push-pull test;
2. In large-ASA patients with secundum ASD (Phase1) (1)The length of ASA >20 mm and bulging >15 mm or a combined total excursion right and left > 15 mm; (2)Secundum ASD with Qp/Qs>1.5 or echocardiographic evidence of right heart enlargement; (3)Failure to cover ASA after trial device-closure of ASD and the unstable device confirmed with push-pull test;
3. Isolated ASA with high risk (Phase2) (1)History of migraine attacks/TIA/cryptogenic stroke without other risks in the last 6 months; (2)Thickening of ASA wall ≥ 5 mm; (3)Spontaneous echo contrast;
4. Left atrial septal pouch (Phase3) (1)History of migraine attacks/TIA/cryptogenic stroke without other risks in the last 6 months; (2)Spontaneous echo contrast in left atrium;

Exclusion Criteria:

1. Acute infection or sepsis;
2. Intra-cardiac thrombus;
3. Carotid, vertebral or basilar artery stenosis > 50% on duplex imaging;
4. Patients unable to grant informed, written consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with effective exclusion of ASA | 12 months
  Assessment of ASA exclusion by echocardiography/MSCT during follow-up. Effective exclusion of ASA was defined as complete coverage of whole ASA.

SECONDARY OUTCOMES:
Procedural or device complications | 12 months
  Procedural or device complications during follow-up
Adverse event rates for all subjects | 12 months
  including migraine (severity, frequency and duration with or without aura), TIA, ischemic stroke or systemic embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Chaowu Yan, PhD and MD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (1):
- Yan Chaowu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No